CLINICAL TRIAL: NCT03491592
Title: Promoting Physical Activity in Latinas Via Interactive Web-based Technology
Brief Title: Web-based Physical Activity Intervention for Latinas
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brown University (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Bess Marcus, Professor of Behavioral and Social Sciences, Brown University School of Public Health, Brown University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R01CA159954 (NIH); R01CA159954 (NIH)
Record Dates: First submitted 2018-03-26; First posted 2018-04-09 (Actual); Last update posted 2023-02-22 (Actual); Status verified 2023-02

CONDITIONS: Inactivity
Keywords: Physical Activity; Latinas; Spanish-language; Text-Message; Exercise; Web-based
MeSH Terms: conditions — Sedentary Behavior; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Enhanced Physical Activity Intervention (Experimental): A data driven enhanced Pasos Hacia La Salud intervention based on results and participant feedback from the motivationally-tailored, Spanish Language, Internet-based Physical Activity intervention in the parent study.
  Interventions: Behavioral: Enhanced Physical Activity Intervention
- Original Physical Activity Intervention (Active Comparator): The original Internet-based program is a computer expert system-driven, individually tailored Spanish language intervention, guided by Social Cognitive Theory (SCT) and the Transtheoretical Model (TTM).
  Interventions: Behavioral: Original Physical Activity Intervention

INTERVENTIONS:
Behavioral: Enhanced Physical Activity Intervention — Participants in the Enhanced Intervention arm will receive all the intervention components of the Original Intervention described above plus: 1) text messages and adaptive goal-setting to drive participants back to the website and keep them there longer, and 2) data-driven, technology supported enhanced intervention content targeting theoretical constructs that influenced PA behavior in Latinas from the parent study.
  Arms: Enhanced Physical Activity Intervention
Behavioral: Original Physical Activity Intervention — Participants in the Original Physical Activity intervention arm of the study will receive the original Spanish language, motivationally-tailored, Internet-based physical activity intervention that specifically addresses the Physical Activity barriers and intervention needs/preferences of Latinas.
  Arms: Original Physical Activity Intervention

SUMMARY:
This renewal builds upon our successful culturally adapted PA intervention for Latinas (Pasos Hacia La Salud, R01CA159954) and expands its focus to the critical area of maintenance of behavior change. This study will test an enhanced version of the original internet intervention in order to achieve greater increases in PA and longer term maintenance. Investigators propose to test this newly developed enhanced intervention (Enhanced Intervention) compared to the original Pasos Hacia La Salud Intervention (Original Intervention) in a 24-month randomized trial (N=300).

DETAILED DESCRIPTION:
In the U.S., Latina women report higher rates of inactivity than their non-Hispanic White and male counterparts, and are disproportionately affected by related health conditions (e.g., cancer, hypertension, heart disease, stroke, diabetes). To address this public health crisis, evidence-based interventions that utilize state-of-the-art technology, theory and methods are needed to increase physical activity (PA) among this high-risk population. Recently, our team conducted a randomized controlled trial (N=205) to test the efficacy of a 6-month culturally adapted, individually tailored, Spanish-language Internet-based PA intervention among Latinas (Pasos Hacia La Salud, R01CA159954) vs. a Wellness Contact Control Internet Group. Increases in minutes/week of moderate-to-vigorous physical activity (MVPA) were significantly greater in the Intervention Group compared to the Control Group at 6 and 12 months (p < .01) but still did not reach levels recommended in the national physical activity guidelines. As improvements in PA in the Intervention Group were significantly associated with website use and increases in self-efficacy, enjoyment, and social support in the parent study, we used these data to inform technology and theory-supported enhancements to the intervention (i.e., text messaging and adaptive goal setting to increase website use and further targeting of the previously mentioned key psychosocial constructs) to achieve even greater increases in PA, and maintain these gains over the long term (24 months) in the renewal of R01CA159954. For the proposed study, 300 Latina women will be randomized to either 1) the original Pasos Hacia La Salud tailored Internet-based PA intervention (Original Intervention) or 2) the data driven, enhanced version of the Pasos Hacia La Salud PA intervention (Enhanced Intervention). We hypothesize that participants in the Enhanced Intervention arm will report significantly more minutes/week of MVPA than participants in the Original Intervention arm at 6 months. We will also examine the maintenance of treatment effects at 12, 18, and 24 months, as well as the costs of delivering the Enhanced vs. Original Intervention programs, and the potential mediators of the intervention-PA relationship. The proposed high reach, low-cost intervention holds great promise in promoting and maintaining the positive health benefits of PA in the lives of Latina women in the United States.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Generally healthy (If asthma and/or high blood pressure, may be able to participate with physician consent)
* Sedentary (Less than 60 minutes per week of moderate or vigorous physical activity)
* Self-identify as Hispanic or Latino (or of a group defined as Hispanic/Latino by the Census Bureau
* Must be able to read and write Spanish fluently
* 18 - 65 years of age
* Daily access to a text-message compatible cell phone and to an Internet-connected device through home, work, or their community

Exclusion Criteria:

* History of coronary heart disease (history of myocardial infarction or symptoms of angina),
* Diabetes that requires insulin and does not have a doctor's approval
* Chronic infectious disease- HIV, Hepatitis C but does not have doctor approval
* Orthopedic conditions which limit mobility, any other serious medical condition that would make PA unsafe (based on modified Physical Activity Readiness Questionnaire)
* Hospitalization due to a psychiatric disorder in the past 3 years
* BMI above 45 kg/m2
* Current or planned pregnancy in the next two year
* Moving from area within two years
* Does not have a cellphone capable of sending and receiving text messages
* Not able to receive materials in the mail, either at your own home or at a mailbox

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 210 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2022-04-01 (Actual); Study Completion 2022-04-01 (Actual)

PRIMARY OUTCOMES:
Change in total weekly minutes of physical activity as measured by an accelerometer | Baseline, 6 months, 12, 18 and 24 months
  For the week prior to each assessment, participants will wear an Actigraph GT3X+ accelerometer which collects min/week of objectively measured MVPA.

CONTACTS AND LOCATIONS:
Locations (1):
- 121 South Main Street, Brown University, Providence, Rhode Island, United States

REFERENCES:
- [Derived] Larsen B, Pekmezi D, Hartman SJ, Dunsiger S, Gilmer T, Groessl E, Marcus B. Costs and Cost-Effectiveness at 12 and 24 Months of an Enhanced Web-Based Physical Activity Intervention for Latina Adults: Secondary Analysis of a Randomized Controlled Trial. J Med Internet Res. 2025 Nov 25;27:e76739. doi: 10.2196/76739. PMID 41289583
- [Derived] Connell Bohlen L, Dunsiger SI, von Ash T, Larsen BA, Pekmezi D, Marquez B, Benitez TJ, Mendoza-Vasconez A, Hartman SJ, Williams DM, Marcus BH. Six-Month Outcomes of a Theory- and Technology-Enhanced Physical Activity Intervention for Latina Women (Pasos Hacia La Salud II): Randomized Controlled Trial. J Med Internet Res. 2024 Jun 6;26:e51708. doi: 10.2196/51708. PMID 38842930
- [Derived] von Ash T, Dunsiger SI, Williams DM, Larsen BA, Bohlen LC, Pekmezi D, Mendoza-Vasconez AS, Benitez TJ, Bock BC, Hartman SJ, Marquez B, Marcus BH. Pasos Hacia La Salud II: A Superiority RCT Utilizing Technology to Promote Physical Activity in Latinas. Am J Prev Med. 2024 Aug;67(2):220-230. doi: 10.1016/j.amepre.2024.03.006. Epub 2024 Mar 13. PMID 38490284
- [Derived] Mendoza-Vasconez AS, Benitez T, Dunsiger S, Gans KM, Hartman SJ, Linke SE, Larsen BA, Pekmezi D, Marcus BH. Pasos Hacia La Salud II: study protocol for a randomized controlled trial of a theory- and technology-enhanced physical activity intervention for Latina women, compared to the original intervention. Trials. 2022 Aug 1;23(1):621. doi: 10.1186/s13063-022-06575-4. PMID 35915473